CLINICAL TRIAL: NCT01792453
Title: MRI Quantification of Gastric and Small Bowel Liquid Volumes Before and After Ingestion of the Standard Oral Solid Delivery 240 mL Water Drink
Brief Title: 240 mL Water Drink Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: University of Michigan (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: A10012013
Record Dates: First submitted 2013-02-13; First posted 2013-02-15 (Estimated); Last update posted 2013-07-04 (Estimated); Status verified 2013-07

CONDITIONS: Healthy
Keywords: Gastrointestinal physiology; MRI; Small bowel water volumes; Gastric volumes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 240 mL water drink (Experimental): Volunteers will be asked to drink 240 mL water drink
  Interventions: Other: Spring water

INTERVENTIONS:
Other: Spring water

SUMMARY:
The GI MRI Research group at the University of Nottingham has been developing new, non-invasive magnetic resonance imaging (MRI) techniques to image the gastrointestinal tract. The investigators now want to characterise; in collaboration with the College of Pharmacy at the University of Michigan, the fasting volumes of gastric and small bowel liquid and their time courses over 2 hours after drinking the FDA recommended 240 mL of water drink for oral solid dosage forms testing.

DETAILED DESCRIPTION:
Solid oral delivery is the most frequently used route of administration for pharmaceutical drug products. Along with other important physiological parameters, the volume of liquid in the small intestine (SILV) has the potential to greatly influence the rate and extent of drug dissolution and absorption in the GI tract, or "oral bioperformance". Modeled small bowel absorption of a drug can vary by more than five-fold as SILV decreases from 500 to 50 ml. To obtain reasonable predictions of oral bioperformance scientists must design meaningful in vitro dissolution tests and mechanistic drug transport models that capture the range of SILV in humans. However, little is known about liquid volumes in the gut, mostly due to invasiveness of previous techniques. A recent study has drawn great attention to the possibility of the liquid in the small intestine existing in discrete liquid "pockets" hence it would also be desirable to monitor the time courses and volumes of individual water pockets in the small intestine.

Magnetic resonance imaging (MRI) is the ideal tool to carry out serial and non-invasive imaging of gastrointestinal function. MRI is inherently suited to image liquid materials and this ability has been exploited to image liquids in the undisturbed gastrointestinal tract. Gastric emptying measurements have been long established and validated. Small bowel liquid volumes measurements have been recently validated against naso-duodenal infusion. Ultimately, the findings with this study will provide novel insights on the volume and distribution of ingested liquids in the gastrointestinal tract.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy; no medical conditions that might affect the study measurements
* Male or female
* Age between 18 and 55 years of age
* Body mass index (BMI) between 18.5 and 24.9 kg m-2
* Suitable for MRI scanning (eg absence of metal implants, infusion pumps and pacemakers as assessed by the MRI safety questionnaire

Exclusion Criteria:

* Previous gastrointestinal surgery (excluding cholecystectomy and appendectomy)
* Known gastrointestinal disease
* Smoking
* History of alcohol or drug abuse
* Taking medication that is likely to affect gastrointestinal function
* Participation in night shift work the week prior to the study day. (Night work is defined as working between midnight and 6 am)
* Strenuous exercise greater than 10 hours per week
* Consumption of more than 21 units of alcohol in a typical week

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2013-02; Primary Completion 2013-03 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Time course of small bowel liquid volume after ingesting 240 mL of water | 0 - 120 mins
  Time course for the volume of freely mobile water in the small bowel over 2 hours

SECONDARY OUTCOMES:
Time course of gastric liquid volume after ingesting 240 mL of water | 0 - 120 mins
  Gastric volumes obtained from MRI as a function of time
Number of liquid pockets in the small bowel | 0 - 120 mins
  Assessment of the number of pockets of liquid in the small bowel as seen on the MR images
Volume of liquid pockets in the small bowel | 0 - 120 mins
  The volume of freely mobile liquid in each of the liquid pockets identified on the MR image
Summary information on the location of liquid pockets by quadrant | 0 - 120 mins
  Details on the distribution of the liquid pockets as seen on the MR images

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Murray, PhD, Principal Investigator — University of Nottingham; Susan Pritchard, MSc, Principal Investigator — University of Nottingham; Caroline Hoad, PhD, Principal Investigator — University of Nottingham; Martin Garnett, Principal Investigator — University of Nottingham; Penny Gowland, PhD, Principal Investigator — University of Nottingham; Robin Spiller, FRCP, Principal Investigator — University of Nottingham; Gregory Amidon, Principal Investigator — University of Michigan; Gordon Amidon, Principal Investigator — University of Michigan; Deanna Mudie, Principal Investigator — University of Michigan; Luca Marciani, PhD, Study Director — University of Nottingham
Locations (1):
- University of Nottingham, Nottingham, Nottingham, United Kingdom